CLINICAL TRIAL: NCT06829108
Title: Association of Transversus Abdominis Plane Block (TAPB) with Postoperative Delirium (POD) in Elderly Patients Undergoing Major Gastrointestinal Surgery: a Retrospective Cohort Study
Brief Title: Association of Transversus Abdominis Plane Block (TAPB) with Postoperative Delirium (POD) in Elderly Patients Undergoing Major Gastrointestinal Surgery
Status: Completed | Type: Observational
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Weidong Mi, Director, Department of Anesthesiology (Cheif expert of National key research and development program of China 2018YFC2001900), Chinese PLA General Hospital
Other Study IDs: PLAGH-TAPB-001
Record Dates: First submitted 2025-02-11; First posted 2025-02-17 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2024-08

CONDITIONS: Regional Anaesthesia; Postoperative Delirium (POD); Transversus Abdominis Plane Block (TAP Block)
Keywords: Regional Anaesthesia; Postoperative Delirium (POD); Transversus abdominis plane block (TAP block)
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- TAPB group and non-TAPB group

SUMMARY:
Postoperative delirium can increase postoperative adverse reactions and prognosis in elderly patients undergoing gastrointestinal surgery. This study studied the effects of ultrasound-guided transversal plane block on postoperative delirium, opioid consumption and prognosis in elderly patients undergoing gastrointestinal surgery, comprehensively evaluated the effectiveness and safety of TAPB, and evaluated its clinical value.

DETAILED DESCRIPTION:
Postoperative delirium (POD) is a common neurocognitive disorder in elderly patients after surgery, which is characterized by attention deficit, memory impairment and confusion, usually occurring within one week after surgery. It occurs in 11%-51% of elderly patients undergoing gastrointestinal surgery and is associated with long-term poor prognosis such as dementia and increased mortality. Risk factors include advanced age, high ASA grade, hypoalbuminemia, and prolonged anesthesia. Regional nerve block (NBs), as the core means of multimodal analgesia, has been shown to reduce the incidence of POD in orthopedic and thoracic surgery by reducing opioid use and stress response, but its effect in elderly gastrointestinal surgery still needs to be further explored. Transverse abdominal muscle plane block (TAPB) is a commonly used technique in abdominal surgery. It can effectively control pain and reduce inflammation and stress response by blocking sensory nerves in the abdominal wall. This study focused on the effect of TAPB on POD in elderly patients undergoing major gastrointestinal surgery, aiming to provide evidence-based evidence for optimizing perioperative anesthesia management.

ELIGIBILITY:
Inclusion Criteria:

1. age ≥65 years;
2. major gastrointestinal surgery, defined as procedures lasting more than one hour and involving partial resection of the stomach or intestines;
3. general anesthesia with endotracheal intubation.

Exclusion Criteria:

1. emergency surgeries;
2. transanal endoscopic microsurgery (TEM);
3. patients with a history of preoperative delirium, altered consciousness, or psychiatric conditions, such as epilepsy, Alzheimer's disease, Parkinson's disease, schizophrenia, and anxiety or depressive disorders, as well as encephalopathies (hepatic, pulmonary, and renal) and hydrocephalus, along with those experiencing significant preoperative visual or auditory impairments;
4. patients who died within 24 h postoperatively or missing data of >50% in their medical records.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: All perioperative data required for this study were obtained from patients at the First Medical Center of the Chinese PLA General Hospital from January 2016 to March 2022.
Sampling Method: Non-Probability Sample
Enrollment: 5220 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2024-10-12 (Actual)

PRIMARY OUTCOMES:
POD incidence within 7 days postoperatively | within 7 days postoperatively

SECONDARY OUTCOMES:
intraoperative sufentanil dosage | intraoperative
length of hospital stay | no more than 1 year
mortality | 30 day after the surgery

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang C, Gao T, Ma HY, Wang R, Sun JJ, Ma LB, Tong L, Fu Q. Association of transversus abdominis plane block (TAPB) with postoperative delirium (POD) in elderly patients undergoing major gastrointestinal surgery: a retrospective cohort study. BMC Anesthesiol. 2025 Sep 29;25(1):464. doi: 10.1186/s12871-025-03363-w. PMID 41023630